CLINICAL TRIAL: NCT03729791
Title: Clinical Trials for Neuroimaging and Electrophysiology in Schizophrenic Patients With Negative Symptoms Using Transcranial Direct Current Stimulation
Brief Title: The Effect of tDCS on Schizophrenia With Negative Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Young Lee, MD, Research Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.001
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; tDCS; negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
  1 arm is active tDCS and 1 arm is sham tDCS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All researchers will conduct research with only the encrypted subject number. A separate third-party researcher will participate to encrypt the subject and adjust the active/sham direction of the tDCS device during the actual research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- actual tDCS (Experimental): 2mA direct current, 20 minutes per session, 2 sessions per day with at least 3hours interval between sessions, a total of 10 tDCS sessions
  Interventions: Device: tDCS
- sham tDCS (Active Comparator): sham direct current, 20 minutes per session, 2 sessions per day with at least 3hours interval between sessions, a total of 10 tDCS sessions
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation (tDCS) is a form of neurostimulation that uses constant, low direct current delivered via electrodes on the head. It can be contrasted with cranial electrotherapy stimulation, which generally uses alternating current the same way

SUMMARY:
The investigators conducted a randomized controlled trial to reveal the effect of tDCS on negative symptoms in patients with schizophrenia and its underlying mechanism using the neuroimaging and electrophysiology.

DETAILED DESCRIPTION:
The project will investigate the use of a novel technique, transcranial direct current stimulation (tDCS) in the treatment of patients with schizophrenia. tDCS permit the application of an extremely weak continuous electrical current to the brain through an anode and a cathode applied on the scalp. Anodal stimulation appears to increase brain activity whereas cathodal stimulation has the opposite effect.

Using anodal and cathodal tDCS the investigators aimed to treat negative symptoms of schizophrenia. The investigators plan to apply tDCS such that it can simultaneously increased activity in the frontal brain areas and reduce activity over temporoparietal cortex, 2 areas involved in the physiopathology of the disease. Real active stimulation will be compare to a sham condition in 44 patients (22 in each group). 44 patients will be included in Seoul National University Hospital

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Schizophrenia
* 1 or more items of Negative symptom score in PANSS > 5

Exclusion Criteria:

* presences of neurological disorder or history
* IQ < 70
* presence of severe personality disorders
* presence of substance use disorder (except nicotin)
* pregnancy
* presence of severe medical condition or disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in psychopathology To assess a patient using PANSS, an approximately 45-minute clinical interview is conducted. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers

SECONDARY OUTCOMES:
The Clinical Assessment Interview for Negative Symptoms (CAINS) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in psychopathology The CAINS is a clinical rating scale for negative symptoms with potent and clear treatment targets for the next generation of pharmacological and psychosocial treatments. It rangs between 0 to 52
Electroencephalography - resting | approximately 2 weeks (baseline and 2 weeks followups)
  changes in lagged phase synchronization and microstate connectivity
Electroencephalography - P300 | approximately 2 weeks (baseline and 2 weeks followups)
  changes in P300
Electroencephalography - MMN | approximately 2 weeks (baseline and 2 weeks followups)
  changes in MMN
Electroencephalography - ERN | approximately 2 weeks (baseline and 2 weeks followups)
  changes in ERN
MRI - grey matter volume | approximately 2 weeks (baseline and 2 weeks followups)
  change in grey matter volume
MRI - cortical thickness | approximately 2 weeks (baseline and 2 weeks followups)
  change in cortical thickness
MRI - cortical surface area | approximately 2 weeks (baseline and 2 weeks followups)
  changes in MRI - cortical thickness
MRI - cortical gyrification | approximately 2 weeks (baseline and 2 weeks followups)
  changes in cortical gyrification
DTI - mean diffusivity (MD) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in MD
DTI - axial diffusivity (AD) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in AD
DTI - radial diffusivity (RD) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in RD
DTI - fractional anisotropy (FA) | approximately 2 weeks (baseline and 2 weeks followups)
  changes in FA
MRI - rsfMRI | approximately 2 weeks (baseline and 2 weeks followups)
  change in BOLD signals
MRI - MRS | approximately 2 weeks (baseline and 2 weeks followups)
  Changes in concentration of N-Acetyl Aspartate, Creatin, Choline, Myoinositol, Glutamate, Glutamine, GABA metabolite concentration change with treatment
fNIRS | approximately 2 weeks (baseline and 2 weeks followups)
  change in level of the Oxy-Hemoglobin
Korean Wechsler Adult Intelligence Scale (K-WAIS) | baseline
  baseline total Intelligence quotient value
Spatial Working Memory | approximately 2 weeks (baseline and 2 weeks followups)
  changes in the spatial working memory ability
California Verbal Learning Test | approximately 2 weeks (baseline and 2 weeks followups)
  changes in verbal learning ability
Letter/Category fluency test | approximately 2 weeks (baseline and 2 weeks followups)
  changes in fluency ability

CONTACTS AND LOCATIONS:
Overall Officials: Tae Young Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No